CLINICAL TRIAL: NCT05763680
Title: Molecular Culture for the Diagnosis of Neonatal Sepsis: Towards Faster Recognition of Uninfected Neonates and Better Antibiotic Stewardship
Brief Title: Molecular Culture for the Diagnosis of Neonatal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jip Groen (Other)
Collaborators: InBiome (Unknown)
Responsible Party: Sponsor-Investigator, Jip Groen, Medical Doctor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: W22_453
Record Dates: First submitted 2023-02-16; First posted 2023-03-10 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Neonatal Sepsis, Early-Onset; Culture Positive Neonatal Sepsis; Culture Negative Neonatal Sepsis; Clinical Sepsis; Microbial Disease; Neonatal Infection; Microbial Colonization; Neonatal Sepsis, Late-Onset
MeSH Terms: conditions — Neonatal Sepsis; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, taken from the umbilical cord postpartum Blood samples, taken peripherally directly following sampling for conventional culture.
  Bacterial swabs, taken from blood sample sites on the umbilical cord to detect possible contaminants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants suspect of neonatal sepsis (early and late onset) up to 90 days postnatally: Infants who are suspect of sepsis, either based on risk factors for infection or on clinical assessment. No restrictions in terms of gestational age
  Interventions: Diagnostic Test: Molecular Culture

INTERVENTIONS:
Diagnostic Test: Molecular Culture — PCR based technique that amplifies the interspace region in bacterial DNA, that is located between the genes coding for 16S and 23S ribosomal subunits. Primers are used for the majority of known pathogenic phyla, i.e. FAFV, Bacteroidetes, Firmicutes and Proteobacteria. The nucleotide length of the Interspace region is species specific for bacterial single species. Bacteria all have one or multiple alleles for this interspace region. The combination of the amount of alleles, as well as the nucleotide strand length, makes for a specific profile that is distinctive for the species. Available software is able to match this profile to a particular pathogen, enabling confirmation and identification of bacteria in samples within 5 hours in our experimental workflow.
  Other Names: IS Pro

SUMMARY:
Rationale: Early diagnosis of sepsis in neonates is complicated as the signs and symptoms are nonspecific. Although blood culture is the gold standard for the diagnosis, false-negative results and long incubation period of 36-72 hours limits the use of blood culture to rule out sepsis at initial suspicion. Since delay in diagnosis may lead to progressive deterioration, antibiotics are often started empirically at initial sepsis suspicion, awaiting results of the blood culture. Consequently, uninfected infants are often unnecessarily exposed to empirical antibiotics. To reduce unnecessary treatment of non-infected infants, an early, sensitive and specific diagnostic tool would be helpful to guide clinicians faster when to discontinue antibiotics. Molecular Culture (MC) via IS-pro is a novel, advanced, molecular culture technique which is able to culture bacteria within 4 hours after blood sampling. MC might thus be a potential diagnostic tool to detect or rule out sepsis in infants quickly, however data on MC for diagnosis of sepsis in this population is limited.

Objective: The aim of this study is to evaluate whether MC is of additive predictive value for the diagnosis sepsis in this vulnerable group.

Study design: Prospective observational cohort study. Study population: All infants suspected for neonatal sepsis of both early and late onset will be eligible for study participation. They will be treated according to the standard local guidelines.

Intervention (if applicable): In case of a suspicion of sepsis at birth, blood will be collected for a conventional blood culture as part of standard care. Additionally, a blood sample will be collected from the umbilical cord for MC.

In case of a suspicion of sepsis not directly postpartum, an additional blood sample will be taken for MC analysis, directly following sampling for conventional culture, implying no extra phlebotomy.

Main study parameters/endpoints: The main study parameter is the discordance in positive and negative outcomes of MC compared to outcomes of conventional blood culture. As the diagnostic accuracy of the conventional blood culture (the current gold standard) is being questioned, the predictive value of MC versus conventional blood culture towards clinical sepsis will also be tested.

DETAILED DESCRIPTION:
Newborns often receive antibiotics for a suspicion of sepsis. Sepsis has high morbidity and mortality in newborns. Around 5% of all newborns and over 85% of very preterm born infants receive antibiotics empirically. Postnatally, antibiotics are often prescribed for presumed bacterial infections on neonatal wards, but in approximately 90-96% of these patients bacterial infection is not proven.

Rapid diagnosis of sepsis in newborns is problematic because clinical signs start subtle and are non-specific. The gold standard for diagnosis of bacterial neonatal sepsis is a conventional blood culture. Unfortunately, bacterial culture is time-consuming (time to result up to 36-72 hours) and lacks sensitivity in this population. For this reason, neonates with risk factors for infection or clinical signs and symptoms of infection are treated with antibiotics empirically at initial sepsis suspicion, awaiting results of the conventional blood culture. Currently more than 85% of very preterm born infants (gestational age <30 weeks) receive antibiotics for the risk of early-onset sepsis in the Netherlands.

There is increasing evidence that, apart from antibiotic resistance, the use of antibiotics in the neonatal period and during childhood alters the microbiome with an increased risk of immediate and long-term adverse effects, such as increased risk for asthma, obesity, allergies and inflammatory bowel diseases (IBD). To avoid unnecessary treatment of non-infected infants, an early, quick, sensitive and specific laboratory test would be helpful to guide clinicians to decide when to discontinue antibiotics as soon as possible.

A promising technique to detect neonatal sepsis quickly and in an earlier stage compared to conventional blood culture is Molecular Culture (MC). MC is an advanced, rapid molecular based culturing technique that is able to identify bacteria within 4 hours after blood sampling. In short, MC is a DNA-based profiling technique, differentiating between bacterial species based on species-specific differences in 16S-23S rDNA interspacer (IS) region nucleotide length by using phylum-specific fluorescently labelled polymerase chain reaction (PCR) primers. A standard IS-pro procedure consists of two separate PCRs. In the first PCR two different primers are added, one primer fluorescently labeling members of the phyla Firmicutes, Actinobacter, Fusobacteria and Verrucomicrobia (FAFV), whereas the second primer labels members of the Bacteroidetes phylum. In the second PCR, a third labeled primer is added targeting members of the phylum Proteobacteria. Subsequently, these PCR products can be amplified and DNA fragments can be separated based on their nucleotide length. Eventually, a typical IS-pro microbial profile will be created, consisting of a set of color-labeled peaks. Each peak representing an individual bacterial operational taxonomic unit (OTU) depending on the nucleotide length of the IS-pro fragment, length of these peaks demonstrating the concentration of this particular OTU, whereas peak colors provides information about the present phyla (FAFV, Bacteroidetes or Proteobacteria). Figure 3 shows a schematic representation of the concept of how the IS-pro procedure works.

Figure 3. Schematic representation of the concept behind the IS-pro procedure. (A) All bacterial species contain at least one IS region in their chromosome. However, many species contain multiple alleles of the IS region. These regions may vary between different alleles. Depicted here is the schematic situation in E. faecalis that contains four alleles of the IS region. Two alleles have a length of 275 nt, and the other two have a length of 377 nt. When amplified, a profile specific for E. faecalis is obtained. (B) IS profiles are highly diverse between different species. The fact that species commonly have multiple alleles with different lengths dramatically increases the differential potential between species. (C) By amplifying IS fragments with phylum-specific fluorescently labeled primers, a next layer of information is added. (D) When an IS profile is made of a sample containing multiple species from different phyla, peaks with different lengths, height, and color are found. These correspond to species, abundance, and phylum. A peak profile may be translated to a list of bacterial species by a software algorithm linked to a database of IS profiles of known bacterial species. The whole IS-pro procedure from unprocessed sample to analyzed data can be performed in 4 h.

In bacterial sepsis, a bacteria has reached the otherwise sterile bloodstream causing sepsis. Both blood culture and MC can detect bacteria and give a positive result (in case a bacteria has been cultured) or a negative result (in case no bacteria was detected). In case the tests are positive, both techniques also show which bacteria was found, which could be used to change antibiotic regimen to target that specific cultured bacteria. However, the process of MC can be finished within 4 hours, which is much shorter than the incubation period of the gold standard blood culture which is 36-72 hours. When there is no sepsis (and thus no bacteria in the bloodstream), the MC will turn out negative also within 4 hours and thus may guide clinicians to stop antibiotics in uninfected infants much faster compared to the conventional blood culture.

Blood cultures are still gold standard, but are generally assumed to have a low sensitivity for the diagnosis of sepsis in newborns and are time consuming. Cases of sepsis may be missed by cultures and a more sensitive diagnostic test such as molecular tests as the MC may be useful. Advances in microbial technology have led to the development of rapid molecular methods, that may be more sensitive than culture. Multiple novel molecular techniques, such as quantitative PCR, broad range conventional PCR and multiplex PCR, have been studied to detect neonatal sepsis. However, these techniques, are directed at specific species which makes it impossible to detect all bacterial species. Thus, anything that is not explicitly searched for will be missed. In contrast, MC had the ability to detect every bacterial species that can cause bacterial neonatal sepsis.

The MC technique has been externally validated to detect bacteria. A series of papers validating all aspects of the MC technique have been published last years. Furthermore, MC is already being used in some hospitals on the intensive care unit to detect bacteria in otherwise sterile specimens like blood, but also on samples obtained from abscesses. In a previous cohort, the investigators from this research group demonstrated that MC may be a useful tool to diagnose sepsis in neonates using cord blood. However, this was a small cohort and no large studies have been performed to analyze the suitability of MC in detecting bacterial sepsis in neonates.

Results from other studies using the MC technique to detect bacteria in human body fluid are promising. In one of these studies 66 samples were collected and tested by conventional culture and MC. In 100% of samples with a positive culture, the MC was also positive. In five samples, the conventional culture turned out to be negative, whereas the MC was positive. The case histories of these five patients were obtained and suggested that the MC findings were highly clinically relevant, and thus may have higher sensitivity compared to conventional blood culture.

In summary, the quick detection makes MC a very promising technique to detect sepsis in newborns using cord blood. However, the suitability of MC in this specific population has not been investigated previously. Therefore, a large, high quality study should be performed to determine the diagnostic accuracy of the MC for sepsis in neonates using cord blood.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age >24 weeks
* Neonates who receive a work up for early onset sepsis (including blood sampling for conventional culture) , either based on risk factors or clinical signs (according to local treatment guidelines) OR
* Infants who receive a work (including blood sampling for conventional culture) up for late onset sepsis

Exclusion Criteria:

* For neonates suspicious of having early onset sepsis: congenital TORCHES infection (Toxoplasma gondii, Rubella virus, Cytomegalovirus, Herpes simplex virus and Treponema pallidum (Syphilis)

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants who are admitted to a clinical ward, either delivery or varying levels of neonatal wards.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of Molecular Culture results to traditional culture | The outcome measure will be assessed after study completion, approximately 2 years after start of inclusion
  Molecular Culture assay will be performed on umbilical cord blood samples and peripherally sampled blood. Results will be compared to conventional peripheral blood cultures that are taken from infants who receive a work up for sepsis.
  Test characteristics, such as sensitivity, specificity, as well as positive and negative predictive values will be given.

SECONDARY OUTCOMES:
Comparison of diagnostic accuracy of Molecular Culture for clinical neonatal sepsis versus conventional peripheral culture | The outcome measure will be assessed after study completion, approximately 2 years after start of inclusion
  Molecular Culture assay results will be used to predict clinical sepsis, compared to conventional peripheral culture.
  Test characteristics, such as sensitivity, specificity, as well as positive and negative predictive values will be given.
  Test characteristics will be given for different definitions of clinical sepsis, given that there is no international consensus on a clinical syndrome definition. Also predictive values of Molecular culture and conventional culture will be calculated for sepsis calculator advice (Kaiser Permanente) as surrogate marker for clinical sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Tim GJ de Meij, MD, PhD, Principal Investigator — Pediatric Gastro-enterologist
Locations (1):
- Maxima Medisch Centrum, Veldhoven, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://inbiome.com/molecular-culture/